CLINICAL TRIAL: NCT00121381
Title: Pimecrolimus Cream 1% Plus Topical Corticosteroid in Patients (2-17 Years of Age) With Severe Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981C2439
Record Dates: First submitted 2005-07-14; First posted 2005-07-21 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic dermatitis; T-cell; pimecrolimus; children; topical corticosteroids
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus 1 % cream plus topical corticosteroid (TCS)
  Interventions: Drug: Pimecrolimus plus topical corticosteroid (TCS)
- 2 (Placebo Comparator): Pimecrolimus vehicle (Placebo) plus topical corticosteroid (TCS)
  Interventions: Drug: Pimecrolimus vehicle (Placebo) plus topical corticosteroid (TCS)

INTERVENTIONS:
Drug: Pimecrolimus plus topical corticosteroid (TCS) — Pimecrolimus 1 % cream plus topical corticosteroid (TCS) twice daily
  Other Names: Elidel
  Arms: 1
Drug: Pimecrolimus vehicle (Placebo) plus topical corticosteroid (TCS) — twice daily administration
  Arms: 2

SUMMARY:
Atopic dermatitis, also called eczema, is characterized by redness, papulation (skin elevation) and pruritus (skin itching). The active ingredient of pimecrolimus inhibits the T-cell activation. These cells are involved in the inflammatory component of the disease. This study will test the safety of pimecrolimus Cream 1% with topical corticosteroid treatment (commonly used in eczema) in patients with severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Severe atopic dermatitis
* 5% of total body surface area (TBSA) affected

Exclusion Criteria:

* Concurrent skin diseases (infections)
* Immunocompromised
* Recently received phototherapy or systemic therapy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400
Dates: Start 2005-05; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events of clinical interest (e.g. skin infections, skin irritation)

SECONDARY OUTCOMES:
Incidence of all other adverse events
Time to relapse of atopic dermatitis
Time to treatment success according to the Investigators Global Assessment (IGA - a measure of disease severity)
Efficacy measured by IGA (treatment success and improvement)
Efficacy measured by improvement in Eczema Area and Severity Index (EASI - a measure of disease severity and extent

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (13):
- United States (13):
  - Pediatric Care Medical Group, Inc., Huntington Beach, California
  - Children's Hospital -San Diego, San Diego, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Dermatology Associates and Research, Coral Gables, Florida
  - Medical College of Georgia - Clinical Investigative Services, Augusta, Georgia
  - Dartmouth Hitchcock Medical Center Section of Dermatology, Lebanon, New Hampshire
  - Wake Forest University School of Medicine Dept. of Dermatology, Winston-Salem, North Carolina
  - Calcagno Research and Development, Gresham, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - 520 Trinity Creek Cove, Cordova, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - A.S.T.H.M.A., Inc, Seattle, Washington